CLINICAL TRIAL: NCT04747314
Title: Proof of Concept Study to Treat Negative Affect in Chronic Low Back Pain
Brief Title: Treating Negative Affect in Low Back Pain Patients
Acronym: TNA-LBP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ajay Wasan, MD, Msc (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Mayo Clinic (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, Ajay Wasan, MD, Msc, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY21010105; UG3AR076568 (NIH)
Record Dates: First submitted 2021-01-06; First posted 2021-02-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low Back Pain; Negative Affectivity
Keywords: chronic pain; low back pain; fibromyalgia; mood; affect; depression; anxiety; opioid use
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Fibromyalgia; Depression; Anxiety Disorders | interventions — Antidepressive Agents; Bupropion; Duloxetine Hydrochloride; Escitalopram; Mirtazapine; Sertraline; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Antidepressant (AD) (Experimental): Subjects will be randomly assigned to receive the antidepressant medication for 4 months under the care of a nurse practitioner and psychiatrist, in addition to their current opioid prescription and weaning guidelines, if applicable. Dosage change and side effects are mitigated by check-in visits (virtually or in-person) every 4 weeks. Non-responders determined at the end of 4 months will be re-randomized to continue receiving AD or EFAR for another 4 months.
  Interventions: Drug: Antidepressant
- Enhanced Fear Avoidance Rehabilitation (EFAR) (Experimental): Subjects will be randomly assigned to receive 8 1-hour physical therapy sessions, pain education, and motivational messaging via Vivify app for 4 months, in addition to their current opioid prescription and weaning guidelines, if applicable. Trained physical/occupational therapists will determine the activities as part of the treatment. Non-responders determined at the end of 4 months will be re-randomized to continue receiving EFAR or AD for another 4 months.
  Interventions: Other: Enhanced Fear Avoidance Rehabilitation
- Antidepressant (AD) + Enhanced Fear Avoidance Rehabilitation (EFAR) (Experimental): Subjects will receive a combination of antidepressant medication and physical therapy for 8 months, in addition to their current opioid prescription and weaning guidelines, if applicable. No re-randomization will be done in this treatment group.
  Interventions: Drug: Antidepressant; Other: Enhanced Fear Avoidance Rehabilitation
- AD -> EFAR (Experimental): Subjects will be randomly assigned to receive the antidepressant medication for 4 months under the care of a nurse practitioner and psychiatrist, in addition to their current opioid prescription and weaning guidelines, if applicable. Dosage change and side effects are mitigated by check-in visits (virtually or in-person) every 4 weeks.
  Non-responders determined at the end of 4 months will be re-randomized to continue receiving AD or EFAR for another 4 months. Those re-randomized to receive EFAR for another 4 months will receive a combination of antidepressant medication and physical therapy, in addition to their current opioid prescription and weaning guidelines, if applicable.
  Interventions: Drug: Antidepressant; Other: Enhanced Fear Avoidance Rehabilitation
- EFAR -> AD (Experimental): Subjects will be randomly assigned to receive 8 1-hour physical therapy sessions, pain education, and motivational messaging via Vivify app for 4 months, in addition to their current opioid prescription and weaning guidelines, if applicable. Trained physical/occupational therapists will determine the activities as part of the treatment.
  Non-responders determined at the end of 4 months will be re-randomized to continue receiving EFAR or AD for another 4 months. Those re-randomized to receive AD for another 4 months will be under the care of a nurse practitioner and psychiatrist, in addition to their current opioid prescription and weaning guidelines, if applicable. Dosage change and side effects are mitigated by check-in visits (virtually or in-person) every 4 weeks.
  Interventions: Drug: Antidepressant; Other: Enhanced Fear Avoidance Rehabilitation

INTERVENTIONS:
Drug: Antidepressant — The antidepressant treatment utilizes antidepressant medication to improve pain, function, and depression outcomes.
  The Antidepressant Treatment History Form (ATHF) will be used to assess adequacy of any prior antidepressant medication treatment and to assist the decision regarding which antidepressant to start. A medication flowchart will help serve as a guideline throughout the drug selection and dosing determination. Weekly assessments completed by subjects will help determine response, tolerability, and necessity for dose adjustment or medication change.
  Other Names: AD: aripiprazole, bupropion, duloxetine, escitalopram, mirtazapine, sertraline, venlafaxine
  Arms: AD -> EFAR; Antidepressant (AD); Antidepressant (AD) + Enhanced Fear Avoidance Rehabilitation (EFAR); EFAR -> AD
Other: Enhanced Fear Avoidance Rehabilitation — The EFAR treatment utilizes physical therapy, pain education, and motivational messaging to improve pain, function, and depression outcomes. Subjects will engage in gradual exposure to exercises and activities they are apprehensive about, such as standing to wash dishes.
  Other Names: EFAR
  Arms: AD -> EFAR; Antidepressant (AD) + Enhanced Fear Avoidance Rehabilitation (EFAR); EFAR -> AD; Enhanced Fear Avoidance Rehabilitation (EFAR)

SUMMARY:
This study will examine how the use of antidepressant, physical therapy, and combination of both affects pain, function, and depression outcomes in chronic low back pain patients.

DETAILED DESCRIPTION:
Approximately 20 million Americans are affected by chronic low back pain and negative affective states such as depression and anxiety. These negative states have all been associated with higher pain intensity, lower pain tolerance, greater use of pain medication, poor pain treatment responses, and higher levels of psychiatric comorbidity among low back pain patients. To improve these outcomes for those who suffer from low back pain, it is important to implement multiple methods with a focus in treating negative affect for pain management rather than using opioids alone.

Antidepressant (AD) and fear avoidance-based physical therapy (EFAR) have individually shown to be promising methods for pain management. In this study, AD, EFAR, and the combination therapy of the two treatments will be explored and implemented to investigate their effectiveness in improving pain, function, depression, and anxiety. The key innovation is testing a new and effective multimodal treatment that can help manage pain, as well as address negative affect.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75
* Pain duration > 6 months
* Must meet the minimum criteria for cognitive function using the PROMIS 2-item cognitive screener (>3)
* Average pain score of > 3/10, with low back pain being the primary pain site
* CLBP meeting Quebec Task Force Classification System categories I-III (from axial pain only to pain radiating beyond the knee without neurological signs). Constant radicular pain associated with sensory loss is highly treatment resistant without surgery
* In the investigator's judgment, evidence of healthcare seeking for low back pain.
* Must meet criteria for high negative affect at 1st study visit: at least 5 on the PHQ-4 (also called the PHQ-2 + GAD-2). Scores above this level are highly associated with having a co-morbid major depression or generalized anxiety disorder diagnosis PHQ-4 scores are used as a proxy for high scores on PROMIS depression and anxiety scales
* Having accessible electronic medical records from UPMC, Brigham and Women's Hospital, or Mayo Clinic, Rochester.
* For those taking opioids (the opioid subgroup), participants must be prescribed opioids currently for at least 3 consecutive months prior to enrollment. Patients must be on opioids for a minimum of three months, taking them on a daily basis or intermittently during the week. The investigators will include those on strong opioids, such as oxycodone and weak opioids, such as tramadol.
* Subject must agree that opioids cannot be increased during the study
* For those taking opioids, no active substance use disorder in the past year as determined by the PI with the use of the Tobacco, Alcohol, Prescription Medications, and Other Substance Tool (TAPS) and a urine toxicology screen. The exceptions are tobacco, medical marijuana use in Pennsylvania or Minnesota, recreational or medical marijuana in the Boston site, or mild prescription opioid use disorder such as opioid misuse
* No acute suicidality or history of major thought disorder (such as mania or psychosis). This will be assessed at study entry which will also include a review of history in EPIC/EMR
* Must possess a mobile device or tablet that can send and receive text messages and access the internet

Exclusion Criteria:

* Back surgery within the past six months
* Active worker's compensation or litigation claims
* New pain and/or psychiatric treatments within 2 weeks of enrollment
* Intent to add new or increase pain treatments during the study period, such as back surgery, nerve block procedures, or medications
* Intent to add new psychiatric treatments during the first 4 months of the study
* Any clinically unstable systemic illness that is judged to interfere with the trial
* History of cardiac, nervous system, or respiratory disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for respiratory depression
* Non-ambulatory status
* Pregnancy or the intent to become pregnant during the study. Women of childbearing potential will all submit a urine sample pregnancy testing at enrollment.
* Not fluent in English and/or not able to complete the questionnaires

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
"Composite Responder", involving the domains of pain, function, and depression. See "Other Pre-Specified Outcomes" for description of these sub-components. | Baseline vs. 4th month of study
  To create the "composite responder" measure, Pain+ function changes will be 1 meaure, and the response rate to depression will be the 2nd component. This is done to simplify the assessment of multi-domain responses. We took this "composite responder" approach since pain, function and depression are inherently related to each other in this patient group with CLBP and high negative affect.
  "Pain+function" and "depression response" will be integrated to determine the "composite responder" rate. A participant could be a pain+function responder, a depression responder, both, or neither. We use standard benchmarks for determining response vs. non-response to each domain. The primary outcome is the rate of response vs. non-response on the "Composite Responder" measure. It will be expressed as percentiles in each category. We will also report the rate of pain+function responders and the rate of depression responders (other pre-specified outcomes).

SECONDARY OUTCOMES:
Change from Baseline Pain Interference at 4 months using PROMIS | Baseline vs. 4 months
  The PROMIS Short Form v1.1 - Pain Interference 4a will assess self-reported consequences of pain with 4 questions ranked on a 5-point scale, from "not at all" to "very much". The minimum raw summed score is 4 and the maximum score is 20. Lower t-scores suggest better outcomes. Outcomes will be measured and compared between the 3 treatment groups.
Change from Baseline Anxiety at 4 months using PROMIS | Baseline vs. 4 months
  The PROMIS Short Form v1.0 - Anxiety 4a will assess self-reported fear, anxious misery, hyperarousal, and somatic symptoms with 4 questions ranked on a 5-point scale, from "never" to "always". The minimum raw summed score is 4 and the maximum score is 20. Lower t-scores suggest better outcomes. Outcomes will be measured and compared between the 3 treatment groups.
Change from Baseline Sleep Disturbance at 4 months using PROMIS | Baseline vs. 4 months
  The PROMIS Short Form v1.0 - Sleep Disturbance 6a self-reported perceptions of sleep quality and sleep depth with 6 questions ranked on a 5-point scale. The minimum raw summed score is 6 and the maximum score is 30. Lower t-scores suggest better outcomes. Outcomes will be measured and compared between the 3 treatment groups.
Change from Baseline Subject's Perception of Change from Treatment at 4 months using Patient Global Impression of Change (PGIC) | Baseline vs. 4 months
  The subject's impression of the impact of the treatment on their pain and function will be measured with a 7-item scale (1 = very much worse, 2 = much worse, 3 = minimally worse, 4 = no change, 5 = minimally improved, 6 = much improved, 7 = very much improved).
Neuropathic pain symptoms change, baseline vs. 4 months | Baseline vs. 4 months
  Using PainDetect, we will compare changes in neuropathic pain symptoms from baseline to 4 months. PainDetect is scored from 0-38 and based on ratings to symptom items scored from '0' (never) to '5' (very strongly).
Fear avoidance beliefs, baseline vs. 4 months | Baseline vs. 4 months
  Using the Fear Avoidance Beliefs Questionnaire, Physical Activities Items, subjects rate from '0' (completely disagree) to '6' (completely agree) four physical activities which may make their pain worse. The items are summed to produce the total score.
Widespread Pain Index | Baseline vs. 4 months
  This measure assesses the degree of widespread pain. 20 body regions are rated by patient as having pain or not. The number of regions is summed to give the total score.
Change in PROMIS Fatigue score from baseline vs. 4 months | Baseline vs. 4 months
  The PROMIS short form v. 1.0 for Fatigue consists of 2 items rated from 1-5, from "not at all" to "very much." The raw score is summed and converted to a T score.

OTHER OUTCOMES:
Change in Physical Function using PROMIS Short Form 2.0. Function is part of the Composite Responder measure, and a pain+function metric more specifically. A subject could be a pain+function responder, a depression responder, both, or neither. | Baseline vs. 4 months
  The PROMIS Short Form v2.0 - Physical Function 6b questionnaire will assess self-reported capability with 6 qualitatively scaled questions ranked on a 5-point scale, from "without any difficulty" to "unable to do" or "not at all" to "cannot do." The minimum raw summed score is 6 and the maximum score is 30. Lower t-scores suggest better outcomes.
Change in Pain Intensity using PROMIS. Pain is part of the Composite Responder measure, and a pain+function metric more specifically. A subject could be a pain+function responder, a depression responder, both, or neither. | Baseline vs. 4 months
  The PROMIS Numeric Rating Scale v1.0 for average pain intensity-- Pain Intensity 1a questionnaire will assess how much a person hurts on average over the past 7 days, with a question ranked on a 11-point scale, from "0 = no pain" to "10 = worst imaginable pain." The minimum raw summed score is 0 and the maximum score is 10. Lower raw response scores suggest lower pain intensity and better outcomes.
Change in Depression using PROMIS. Depression is part of the "Composite Responder" measure. A subject could be a pain+function responder, a depression responder, both, or neither. | Baseline vs. 4 months
  The PROMIS Short Form v1.0 - Depression 4a will assess self-reported negative mood and views of self with 4 questions ranked on a 5-point scale, from "never" to "always". The minimum raw summed score is 4 and the maximum score is 20. Lower t-scores suggest better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Wasan, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - BWH Pain Management Center, Chestnut Hill, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - UPMC Pain Medicine At Centre Commons, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wasan AD, Edwards RR, Kraemer KL, Jeong J, Kenney M, Luong K, Cornelius MC, Mickles C, Dharmaraj B, Sharif E, Stoltenberg A, Emerick T, Karp JF, Bair MJ, George SZ, Hooten WM. Back Pain Consortium (BACPAC): Protocol and Pilot Study Results for a Randomized Comparative-Effectiveness Trial of Antidepressants, Fear Avoidance Rehabilitation, or the Combination for Chronic Low Back Pain and Comorbid High Negative Affect. Pain Med. 2023 Aug 4;24(Suppl 1):S105-S114. doi: 10.1093/pm/pnad006. PMID 36715655

DOCUMENTS (1):
  • Informed Consent Form (2024-09-03): https://cdn.clinicaltrials.gov/large-docs/14/NCT04747314/ICF_000.pdf